CLINICAL TRIAL: NCT06770153
Title: Comparison Between the Use of the Tensioner and Standard Surgical Technique for Ligament Balancing of Total Knee Prostheses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TKA-BALANCE
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Knee Injuries
Keywords: Knee prosthesis; prosthesis; knee
MeSH Terms: conditions — Knee Injuries | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator)
  Interventions: Procedure: standard
- Tensor (Experimental)
  Interventions: Procedure: Tensor

INTERVENTIONS:
Procedure: Tensor — balancing will be carried out using the TEMIS DePuy tensioner and carrying out any releases according to the gap-balancing technique
  Arms: Tensor
Procedure: standard — primary TKA implantation with ligament balancing without use of the tensioner
  Arms: Standard

SUMMARY:
the objective of the present study is to compare the post-operative laxity using stress radiographs and clinical scores in two groups of patients undergoing primary PS TKA with identical prosthetic model performed in two specialized centers, of which one group implanted with standard technique and one group through the intraoperative use of the tensioner

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects candidates for primary cemented total knee prosthesis model Attune PS mobile plate DePuy.
* Patients who possess all the psychophysical capabilities to be able to undergo the operation and all the check-ups with radiological tests included (e.g. all patients who are not willing to go to the institute for all the scheduled follow-up visits will be excluded) .
* Patients who have signed the "informed consent" approved by the Ethics Committee.
* Patients who are aged between 50-85.

Exclusion Criteria:

* Social conditions that prevent participation in the study in all its phases (homeless patients, with restrictions on personal freedom, etc.)
* Patients suffering from deep venous insufficiency of the lower extremities or with a personal or family history of deep venous thrombosis or pulmonary embolism
* Patients with a history of erysipelas in the lower extremities
* Patients suffering from neurological or psycho-cognitive disorders
* Patients suffering from post-traumatic arthrosis
* Patients who have already undergone prosthetic surgery and/or arthrodesis at the level of a lower limb joint
* Patients with axial knee deformities >15°
* Pregnant female patients
* Patients with rheumatic diseases

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
radiographical images | at baseline, after 3 months, after 6 months anfer 12 months
  take stress x-rays (150 N) of the knee using TELOS to objectively and reproducibly analyze the lift-off (distance between the prosthetic component femoral and the tibial prosthetic component measured in mm)

SECONDARY OUTCOMES:
Hip-Knee-Anke Angle | at baseline, after 3 months, after 6 months anfer 12 months
  Hip-Knee-Anke Angle (HKA) on orthostatic panoramic radiographs of the pre- and post-operative lower limbs of the knee.
Visual Analogue Scale | at baseline, after 3 months, after 6 months anfer 12 months
  Visual Analogue Scale (VAS) for pain: a scale from 0 to 10 where 0 is no pain and 10 is the worst pain ever

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided